CLINICAL TRIAL: NCT03082014
Title: EffecTs of Amlodipine and Other Blood PREssure Lowering Agents on Microvascular FuncTion in Small Vessel Diseases
Brief Title: Effects of Amlodipine and Other Blood Pressure Lowering Agents on Microvascular Function
Acronym: TREAT-SVDs
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: completed for the primary study group of sporadic SVD patients, halted prematurely for the additional study group due to slow recruitment at 26 of 30 CADASIL patients in December 2022
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: University of Edinburgh (Other); Maastricht University Medical Center (Other); UMC Utrecht (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Martin Dichgans, Prof. Dr. Martin Dichgans, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TRE-1486--0105-I
Record Dates: First submitted 2017-03-08; First posted 2017-03-17 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: Hypertension; Cerebrovascular Reactivity; Blood Pressure Variability
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Hypertension | interventions — Amlodipine; Losartan; Atenolol

STUDY DESIGN:
Intervention Model Description: TREAT-SVDs is a multi-centre, multinational phase III b clinical trial with a three sequence crossover design. It will be carried out as a rater blinded trial which is also known as PROBE-design (prospective, randomised, open-label trial with blinded endpoint assessment).
Who Masked: Outcomes Assessor
Masking Description: Cerebrovascular reactivity measures will be assessed centrally by a blinded rater.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Active Comparator): Amlodipine for 4 weeks, Losartan for 4 weeks, Atenolol for 4 weeks.
  Interventions: Drug: Amlodipine; Drug: Losartan; Drug: Atenolol
- Arm B (Active Comparator): Atenolol for 4 weeks, Amlodipine for 4 weeks, Losartan for 4 weeks.
  Interventions: Drug: Amlodipine; Drug: Losartan; Drug: Atenolol
- Arm C (Active Comparator): Losartan for 4 weeks, Atenolol for 4 weeks, Amlodipine for 4 weeks.
  Interventions: Drug: Amlodipine; Drug: Losartan; Drug: Atenolol

INTERVENTIONS:
Drug: Amlodipine — blood pressure lowering agent - dihydropyridine Ca2+-channel blocker
Drug: Losartan — blood pressure lowering agent - angiotensin-receptor blockers
Drug: Atenolol — blood pressure lowering agent - beta-blocker

SUMMARY:
Multicentre, multinational, prospective randomised, open-label, 3 sequence crossover phase III b clinical trial with blinded endpoint assessment (PROBE-design)

* in 75 patients with sporadic small vessel diseases (SVDs) and
* in 30 patients with cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL)

DETAILED DESCRIPTION:
TREAT-SVDs will be carried out as a multicentre open label trial at five trial sites across 3 European countries: Germany, the Netherlands, and the United Kingdom.

Patients meeting eligibility criteria will be randomly allocated to one of three sequences of antihypertensive treatment which are given as open-label oral medications in standard dose in the following order

Arm A: Amlodipine > Losartan > Atenolol

Arm B: Atenolol > Amlodipine > Losartan

Arm C: Losartan > Atenolol > Amlodipine.

The study starts with a two week run-in phase. During these first two weeks, patients are not allowed to take antihypertensive drugs except for the rescue medication. After the run-in period,every patient will take subsequently three different antihypertensive drugs (each drug from a separate drug class) according to the randomly assigned arm. Each study drug will be administered for four weeks.

Patients will be monitored telemetrically with a dedicated BP device during the whole trial period of 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients may be enrolled in the trial if all of the following criteria have been met:

* Symptomatic SVD defined as

  * History of clinical lacunar stroke in the last 5 years with a corresponding small subcortical infarct visible on MRI scan or CT scan* compatible with the clinical syndrome.

    *On MRI, recent infarct is defined as a diffusion-weighted imaging (DWI) lesion on the acute MRI scan. On CT, recent infarct is defined as a novel infarct on CT within 3 weeks after the event that was not visible on the admission CT. Patients admitted to the hospital with an obvious lacunar syndrome and an admission CT/CT perfusion compatible with a lacunar infarct but without an MRI in the (sub)acute stage and no repeat CT performed in the context of clinical care can be recruited for TREAT-SVDs. After providing informed consent they will be invited for the screening visit including a 3T MRI. The 3T MRI will be used to verify the presence of a new lesion, relative to the admission CT, compatible with a lacunar infarct and compatible with the lacunar syndrome. If such a lesion is present the patient will undergo the further TREAT-SVDs workup. If no such lesion is observed the patient will be excluded from the study and considered as a screening failure.
  * or cognitive impairment defined as visiting a memory clinic with cognitive complaints, objective cognitive impairment*, and capacity to consent, and with confluent deep white matter hyperintensities (WMH) on MRI (defined on the Fazekas scale as deep WMH score ≥ 2)

    *concluded by the treating physician based on a validated cognitive measurement tool (for example but not limited to MoCA or CAMCOG)
  * or a diagnosis of CADASIL established by molecular genetic testing of the NOTCH3 gene (presence of an archetypical, cysteine-affecting mutation) or the presence of granular osmiophilic material in ultrastructural, electron microscopy analysis of skin biopsy
* Indication for antihypertensive treatment (as defined by meeting one of the following):

  * Hypertension defined as SBP ≥ 140 mmHg or diastolic BP (DBP) ≥ 90 mmHg without antihypertensive treatment or use of an antihypertensive drug for previously diagnosed hypertension
  * Prior history of stroke or transient ischaemic attack (TIA)
* Age 18 years or older
* Written informed consent

Exclusion Criteria:

Patients will be excluded from the trial for any of the following reasons:

* Inclusion criteria are not met
* Unwillingness or inability to give written consent
* Pregnant or breastfeeding women, women of childbearing age not taking contraception.

Acceptable contraception in women of childbearing age is a "highly effective" contraceptive measure as defined by the Clinical Trials Facilitation Group and includes combined (oestrogen and progesterone containing) or progesterone-only contraception associated with inhibition of ovulation, or intrauterine device, or bilateral tubal occlusion.

* Contraindications to MRI (pacemaker, aneurysm clip, cochlear implant etc.)
* Other major neurological or psychiatric conditions affecting the brain and interfering with the trial design (e.g. multiple sclerosis)
* In case of clinical lacunar stroke syndrome other causes of stroke such as

  * ≥ 50% luminal stenosis (NASCET) in large arteries supplying the area of ischaemia
  * major-risk cardioembolic source of embolism (permanent or paroxysmal atrial fibrillation, sustained atrial flutter, intracardiac thrombus, prosthetic cardiac valve, atrial myxoma or other cardiac tumours, mitral stenosis, recent (< 4 weeks) myocardial infarction, left ventricular ejection fraction less than 30%, valvular vegetations, or infective endocarditis)
  * other specific causes of stroke identified (e.g. arteritis, dissection, migraine/vasospasm, drug misuse)
* Other stroke risk factor requiring immediate intervention that would preclude involvement in the trial
* Renal impairment (eGFR < 35ml/min)
* Life expectancy < 2 years
* Use of > 2 antihypertensive drugs at maximum dose or equivalent (one drug at the maximum dose and two drugs at half of the maximum dose) for an appropriate BP control
* Contraindications to the applied antihypertensive drugs as known

  * Severe aortic stenosis
  * Bilateral renal artery stenosis
  * Severe arterial circulatory disorders
  * Atrioventricular block II° or III° or sick sinus syndrome
  * Heart failure (NYHA III or IV)
  * Bradycardia, resting heart rate < 50/min
  * Bronchospastic diseases such as severe bronchial asthma
  * Severe hepatic dysfunction such as liver cirrhosis
  * Use of monoamine oxidase (MAO)-A-blockers
  * Use of simvastatin > 20mg/d
  * Metabolic acidosis
  * Disturbed electrolyte homeostasis such as hypercalcaemia, hypokalaemia, and hyponatraemia
  * Symptomatic hyperuricaemia (gout)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Cerebrovascular Reactivity (CVR) at 4 weeks of Monotherapy | baseline measure at the end of the run-in phase (week 2); after 4 weeks of each monotherapy (week 6, week 10, and week 14)
  The primary outcome variable is CVR as determined by blood oxygen level-dependent (BOLD) MRI (T2*) brain scan response to hypercapnic challenge at the end of the 2 week run-in phase and after 4 weeks of monotherapy while still on medication.

SECONDARY OUTCOMES:
Change from Baseline Mean Systolic Blood Pressure (SBP) at the last week of each treatment phase | within the last week of the run-in phase and within the last week of each treatment phase
  Mean SBP assessed by daily telemetric monitoring within the last week of the run-in phase and within the last week of each treatment phase
Change from Baseline Blood Pressure Variability (BPv) at the last week of each treatment phase | within the last week of the run-in phase and within the last week of each treatment phase
  BPv operationalized as coefficient of variation (100*std/mean SBP) across multiple measurements and assessed by daily telemetric monitoring within the last week of the run-in phase and within the last week of each treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dichgans, Prof., Study Director — Institute for Stroke and Dementia Research; Joanna Wardlaw, Prof., Principal Investigator — Neuroimaging Sciences and Brain Research Imaging Centre; Robert van Oostenbrugge, Prof., Principal Investigator — Maastricht University Medical Center (UM), Department of Neurology; Geert Jan Biessels, Prof., Principal Investigator — UMC Utrecht Brain Center Robert Magnus (UMCU); Peter Rothwell, Prof., Principal Investigator — Nuffield Department of Clinical Neurosciences, Oxford (UOXF)
Locations (5):
- Insitute for Stroke and Dementia Research, Munich, Germany
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - University Medical Center Utrecht, Utrecht
- United Kingdom (2):
  - Nuffield Department of Clinical Neurosciences, Oxford, England
  - Centre for Clinical Brain Sciences, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kopczak A, Stringer MS, van den Brink H, Kerkhofs D, Blair GW, van Dinther M, Reyes CA, Garcia DJ, Onkenhout L, Wartolowska KA, Thrippleton MJ, Kampaite A, Duering M, Staals J, Lesnik-Oberstein S, Muir KW, Middeke M, Norrving B, Bousser MG, Mansmann U, Rothwell PM, Doubal FN, van Oostenbrugge R, Biessels GJ, Webb AJS, Wardlaw JM, Dichgans M; TREAT-SVDs collaborators. Effect of blood pressure-lowering agents on microvascular function in people with small vessel diseases (TREAT-SVDs): a multicentre, open-label, randomised, crossover trial. Lancet Neurol. 2023 Nov;22(11):991-1004. doi: 10.1016/S1474-4422(23)00293-4. PMID 37863608
- [Derived] Kopczak A, S Stringer M, van den Brink H, Kerkhofs D, W Blair G, van Dinther M, Onkenhout L, A Wartolowska K, Thrippleton MJ, Duering M, Staals J, Middeke M, Andre E, Norrving B, Bousser MG, Mansmann U, Rothwell PM, N Doubal F, van Oostenbrugge R, Biessels GJ, Webb AJ, Wardlaw JM, Dichgans M. The EffecTs of Amlodipine and other Blood PREssure Lowering Agents on Microvascular FuncTion in Small Vessel Diseases (TREAT-SVDs) trial: Study protocol for a randomised crossover trial. Eur Stroke J. 2023 Mar;8(1):387-397. doi: 10.1177/23969873221143570. Epub 2022 Dec 16. PMID 37021189